CLINICAL TRIAL: NCT03766659
Title: Endoscopic Ultrasound-guided Fine Needle Biopsy With Macroscopic On-Site Evaluation vs Fine Needle Aspiration With Rapid On-Site Evaluation for Solid Pancreatic Lesions: A Multi-centered Prospective Randomized Controlled Trial (MORE Trial)
Brief Title: EUS-FNB With MOSE vs EUS-FNA With ROSE
Acronym: MORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MORE
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: International multicenter prospective randomized comparative study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOSE (Other): EUS-FNB with MOSE
  Interventions: Diagnostic Test: MOSE
- ROSE (Other): EUS-FNA with ROSE
  Interventions: Diagnostic Test: ROSE

INTERVENTIONS:
Diagnostic Test: MOSE — EUS-FNB with MOSE
  Arms: MOSE
Diagnostic Test: ROSE — EUS-FNA with ROSE
  Arms: ROSE

SUMMARY:
Endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) is an indispensable tool for tissue acquisition for pancreatic lesions. However, FNA alone has several limitations including inadequate acquisition of cells, and unable to provide core tissue for further histological analysis. The use of rapid on-site evaluation (ROSE) by cytopathologist has the biggest impact on improving diagnostic accuracy and is regarded as the gold standard for EUS-FNA. Unfortunately, it is not widely available due to limited resources.

In order to overcome these limitations, new fine needle biopsy (FNB) needles have been recently developed to collect not only cells but also the entire core tissue for histological analysis. Having core biopsy with preserved tissue provides additional advantages of allowing molecular analysis, which are of emerging importance in cancer management. Early results comparing FNB with FNA showed the superiority of FNB over FNA in the absence of ROSE. Data comparing FNB and FNA with ROSE are limited. In order to study to true merits of FNB over FNA, comparison with the most optimal method is necessary.

DETAILED DESCRIPTION:
The purpose of this study is to compare the diagnostic yield of EUS-FNB with MOSE vs EUS-FNA with ROSE.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* Referred for EUS-guided tissue acquisition of solid pancreatic lesions greater than 1cm in the largest diameter

Exclusion Criteria:

* Coagulopathy
* Altered anatomy
* Contraindications for conscious sedation
* Pregnancy
* Those who cannot provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 1 month after Procedure
  the proportion of patients with adequate tissue for diagnosis

SECONDARY OUTCOMES:
morbidity rate | 1 month after Procedure
  Procedure-related morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery; The Chinese University of Hong Kong, Hong Kong, Hong Kong